CLINICAL TRIAL: NCT05939908
Title: To Assess Prevalence of Sarcopenia Using Hand Grip Strength (HGS) as a Marker in Patients With T2DM
Brief Title: Assessment of Hand Grip Strength Using Jamar Dynamometer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diabetes Foundation, India (Other)
Collaborators: National Diabetes Obesity and Cholesterol Foundation (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Other Study IDs: HGS
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Type2diabetes
MeSH Terms: interventions — Hand Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Using Jamar Dynamometer for Grip Strength. — Hand grip strength as a marker by using JAMAR hand grip dynamometer in patients with T2DM.

SUMMARY:
Hand grip strength will be measured for all the type 2 diabetic patients. Measurement of maximal grip strength will be performed using Jamar dynamometers, which estimate the muscle strength primarily generated by the flexor muscles of the hand and the forearm. The Jamar displays grip force in both pounds and kilograms, with a maximum of 200 lb (90 kg). It has a peak-hold needle that automatically retains the highest reading until reset. The Jamar test is isometric, with no perceptible motion of the handle, regardless of the grip strength applied. The participants will be encouraged to produce their maximal grip strength. Three trials will be recorded, consisting of a 2-4-second maximal contraction, with a 30-second rest period between each trial. The average of the three readings will be taken.

DETAILED DESCRIPTION:
Sarcopenia is an age related, progressive, and generalized skeletal muscle disorder involving the accelerated loss of muscle mass and function and physical performance below a defined threshold1. It is associated with increased adverse outcomes including increased risk falls, physical frailty, prolonged hospitalization, dependency, physical disability and impairment, limitation of mobility, decreased quality of life and increased mortality. Sarcopenia is known to be more prevalent in older populations, but the decline in muscle mass starts from ~40 years onwards2.

Sarcopenia not only affects the ability to lead an active lifestyle but also contributes to increased obesity, type 2 diabetes (T2DM) reduced quality of life, osteoporosis, and metabolic health1.

Hand grip strength (HGS) is considered as an important value when diagnosing sarcopenia. Lower muscle strength using HGS is mandatory to diagnose sarcopenia. EWGSOP group recommends that the mean reference cut-off value of hand grip is < 30 kg in men and < 20 kg in women.

There is evidence that strength could be an important risk factor for diabetes. Low hand-grip strength has been predictive of incident diabetes in prospective cohort studies3. Lower grip strength was associated with higher prevalence of diabetes, independent of confounding factors, across all ethnicities in both men and women. Diabetes prevalence was approximately three- to fourfold higher in South Asian participants across all levels of grip strength3 .

However, there are no studies in India assessing sarcopenia in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

All patients with Type 2 diabetes of any duration coming for first time in OPD

Exclusion Criteria:

1. Patients with hand fracture
2. Thyroid dysfunction
3. Any musculoskeletal condition causing difficulty in holding the dynamometer
4. Patients with type1 diabetes (T1DM) and gestational diabetes (GDM)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: T2DM patient visiting Fortis CDOC Hospital and meeting the Inclusion Criteria will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of age and gender specific prevalence of sarcopenia using HGS in patients with T2DM | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — Fortis CDOC Hospital
Locations (1):
- Fortis CDOC Hospital, Delhi, India

IPD SHARING:
Plan to Share IPD: No